CLINICAL TRIAL: NCT04052659
Title: A Study to Evaluate the Efficacy and Safety of Sintilimab (IBI308) in Combination With Chidamide and Azacitidine in the Refractory or Relapsed PTCL: A Phase 2, Single-center, Single-arm, Open Label Trial
Brief Title: Sintilimab (IBI308) in Combination With Chidamide and Azacitidine in Refractory or Relapsed PTCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jun Zhu, Principal Investigator, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI308Y016
Record Dates: First submitted 2019-08-09; First posted 2019-08-12 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — sintilimab; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (sintilimab,chidamide and azacitidine) (Experimental): Sintilimab: 200 mg IV, Q3W, d1
  Chidamid: 30 mg PO, BIW, d1, d4
  Azacidine: 100 mg SC, Q3W, d1-7
  Interventions: Drug: Sintilimab; Drug: Chidamide; Drug: Azacidine

INTERVENTIONS:
Drug: Sintilimab — 200 mg IV, every 3 weeks, d1
  Other Names: IBI308
Drug: Chidamide — 30 mg PO, 2 times every week, d1 and d4
  Other Names: Epidaza
Drug: Azacidine — 100 mg SC, every 3 weeks, d1 to d7
  Other Names: Ladakamycin

SUMMARY:
This is a single-arm, single-center Phase II clinical trial for patients with relapsed or refractory Peripheral T-cell lymphoma (PTCL). Immunotherapy with anti-PD-1 antibodies, such as sintilimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chidamide and azacitidine may respectively stop the growth of tumor cells by blocking histone deacetylation and DNA methylation enzymes needed for cell growth. Giving chidamide and azacitidine with sintilimab these three drugs may work better than single drug or combination of two drugs in treating patients with relapsed or refractory peripheral T-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

To determine the objective response rate (ORR).

SECONDARY OBJECTIVES:

1. To determine the complete response rate (CRR).
2. To determine the duration of response (DOR).
3. To determine the progression free survival (PFS).
4. To determine the overall survival (OS).
5. To determine the safety.

EXPLORATORY OBJECTIVES:

Assess the correlation between the expression of PD-L1, CD4, CD8, CD68 in tumor microenvironment and the efficacy of combined therapy in relapsed or refractory peripheral T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed PTCL;
* Disease status defined as relapsed or refractory after >=1 prior treatment lines;
* Prior use of HDACi or PD-1/PD-L1 antibodies or demethylation drugs is allowed;
* At least one measurable disease (defined as ≥ 1.5 cm in length-diameter, or 1.1~1.5 cm in length-diameter and >1.0 cm in short-diameter ) ；
* ECOG PS 0~2；
* Provide written informed consent for the trial；
* 18 ≤ age ≤ 80；
* Life expectancy ≥12 weeks;
* Adequate organ and bone marrow function, laboratory tests should be received within 7 days prior to the use of the research drug and meet the eligibility requirements;
* Subjects of reproductive potential must be willing to use adequate contraception during the course of the study and through 120 days after the last dose of study medication.

Exclusion Criteria:

* Known central nervous system lymphoma or cutaneous T-cell lymphoma;
* Received any immunesuppressive drugs within 4 weeks of the first dose of study medicationy, not including topical corticosteroids or systemic corticosteroids in physiological doses (≤10 mg/day prednisone or equivalent dose of other steroid);
* Patients with active autoimmune diseases requiring systematic treatment in the past two years;
* Received or plan to receive any attenuated vaccines within 4 weeks of the first dose of study medication;
* Received the last anti-tumor therapy within 4 weeks of the first dose of study medication or have not recovered (recovery defined as baseline or ≤ grade 1) from adverse events due to anti-cancer agents;
* Currently participating in an interventional clinical study, unless participating in observational study or during follow-up period of an interventional study;
* Received any investigational agent within 4 weeks of the first dose of study medication;
* Subjects with interstitial lung disease or lung disease that may interfere with the detection or treatment of suspected drug-related pulmonary toxicity;
* Other primary malignancy;
* Known history of allogeneic organ or allogeneic hemopoietic stem cell transplantation;
* Received autologous hemopoietic stem cell transplantation within 90 days of the first dose of study medication;
* Received major surgery or unhealed wound, ulcer or fracture within 4 weeks of the first dose of study medication;
* Active tuberculosis；
* Known primary immunodeficiency；
* Known allergy or hypersensitivity to any monoclonal antibodies or any components used in their preparation;
* Uncontrolled concomitant disease;
* Patients with active hepatitis. Patients who are positive for hepatitis B Surface Antigen (HBsAg) or hepatitis C Virus (HCV) antibodies at screening stage must pass further detection of hepatitis B Virus (HBV) DNA titer (no more than 50 IU/mL) and HCV RNA (no more than the lower limit of the detection method);
* History of gastrointestinal perforation and /or fistula within 6 months before enrollment;
* Hemophagocytic syndrome；
* Uncontrolled third space effusion, e.g. ascites or pleural effusion cannot be drained or controlled;
* Women who are pregnant or nursing；
* According to the researchers' judgment, patients' underlying condition may increase their risk of receiving research drug treatment, or confuse their judgment on toxic reactions;
* Other researchers consider it unsuitable for patients to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-15 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) by Lugano 2014 up to 24 months | Up to 24 months
  Proportion of subjects who achieve complete response (CR) or partial response (PR) by Lugano 2014 response criteria

SECONDARY OUTCOMES:
Complete remission rate (CRR) by Lugano 2014 up to 24 months | Up to 24 months
  Proportion of subjects who achieve complete response (CR) by Lugano 2014 response criteria
Duration of response (DOR) up to 24 months | Up to 24 months
  DOR is defined as the time from the date of first remission to the date of disease progression or death whichever is earlier
Progression free survival (PFS) up to 24 months | Up to 24 months
  PFS is defined as the time from the treatment date to the date of disease progression per the Lugano 2014 Response Criteria or death regardless of cause
Overall survival (OS) up to 24 months | Up to 24 months
  OS is defined as the time from treatment to the date of death
Incidence and Severity of adverse events by CTCAE v5.0 up to 90 days post-treatment | Up to 90 days post-treatment
  Incidence and Severity of adverse events as assessed by CTCAE v5.0

OTHER OUTCOMES:
Identification of potential biomarkers predictive of response to treatment | Up to 24 months
  The correlation of clinical response with the expression of PD-L1, CD4, CD8, CD68 in tumor environment

CONTACTS AND LOCATIONS:
Overall Officials: Yuqin Song, Doctor, Principal Investigator — Cancer Hospital of Beijing University
Locations (1):
- Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No